CLINICAL TRIAL: NCT06534957
Title: Online Mindfulness-based Stress Reduction Intervention for Patients With Breast Cancer Receiving Chemotherapy
Brief Title: Online Mindfulness-based Stress Reduction for Patients Receiving Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medicos e Investigadores en la Lucha contra el Cancer de Mama (Other)
Responsible Party: Principal Investigator, Fernanda Mesa-Chavez, Principal Investigator, Medicos e Investigadores en la Lucha contra el Cancer de Mama
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECA-MIND-QT
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Stress
Keywords: mindfulness-based stress reduction; chemotherapy-related stress; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Given the nature of the intervention, the study will be open and participants will know which group they were randomized to. However, the study will be blinded to the statistician in order to reduce the risk of introducing bias when interpreting the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be assessed with the study surveys at baseline (T1), will participate in the online MBSR intervention for the next 6 weeks, and will be subsequently reassessed with the study surveys at 7 weeks (T2) and at 11 weeks (T3) of follow-up.
  Interventions: Other: Online mindfulness-based stress reduction
- Wait-list control group (No Intervention): A wait-list control group will be used with the objective that all participants have the opportunity of receiving the online MBSR intervention and at the same time allow comparison of the effectiveness of the program with a group without intervention. Given that treatment-related stress has an important negative impact on patients' wellbeing, it is appropriate to offer the control group the possibility of receiving the intervention if its effectiveness is demonstrated.
  The control group will be assessed with the study surveys at baseline (T1), will not participate in the online MBSR intervention for the next 6 weeks, and will be subsequently reassessed with the study surveys at the same timepoints as the intervention group at 7 weeks (T2) and at 11 weeks (T3) of follow-up. Upon completion of recruitment and follow-up of all participants, the study will end, and the control group will be able to receive the online MBSR intervention according to their preference.

INTERVENTIONS:
Other: Online mindfulness-based stress reduction — The online MBSR intervention sessions will be available in a website created specifically for this purpose, where each pre-recorded session will be uploaded so that each patient can begin the intervention at the same time as their chemotherapy regimen. Each session will last approximately 1 hour, for a total of 6 sessions. The topics that will be covered in these sessions include: mindfulness overview, stress and suffering, emotional regulation, meditation, management of stressful situations, self-compassion and acceptance. Participants will watch 1 session per week following the order that will be indicated on the website; patients will be encouraged to watch the sessions during their chemotherapy infusions. During these sessions, patients will be instructed in mindfulness practice and will perform targeted exercises to promote complete consciousness, including mindful body awareness (body scan), gentle yoga exercises, and meditation.
  Arms: Intervention group

SUMMARY:
The goal of this prospective, waitlist-controlled, 1:1 randomized study is to evaluate if an online mindfulness-based stress reduction (MBSR) intervention reduces treatment-related stress levels among patients with breast cancer receiving chemotherapy.

The main questions it aims to answer are:

* Does an online MBSR intervention reduce stress levels (measured through the Perceived Stress Scale) among participants?
* Does an online MBSR intervention reduce anxiety, depression, insomnia, fatigue, nausea, diarrhea, constipation, pain, and peripheral neuropathy (measured through the PRO-CTCAE of the National Cancer Institute) among participants?

Researchers will compare the online MBSR intervention to no intervention to see if online MBSR reduces treatment-related stress.

Participants will:

* Participate in an online MBSR intervention or no intervention for 6 weeks
* Answer the study surveys at baseline, 7 weeks, and 11 weeks of follow-up

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age ≥18 years
* Diagnosis of non-metastatic breast cancer
* Plan to start neoadjuvant or adjuvant chemotherapy in <4 weeks
* Internet access at home or in their mobile phone
* Availability to participate in the online MBSR intervention for 6 weeks
* Availability to answer the study surveys
* Provision of signed informed consent

Exclusion Criteria:

* Disease recurrence
* Current meditation or mindfulness practice
* Inability to read or write

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Stress | 11 weeks
  Measured through the Perceived Stress Scale (PSS). The PSS is a self-report instrument that assesses the level of perceived stress over the past month. It consists of 10 items that are rated using a 5-point Likert scale (0: Never; 1: Almost never; 2: Sometimes; 3: Fairly often; 4: Very often). The total score is obtained by adding the scores of the 10 items, obtaining a total value between 0-40, where higher scores indicate a higher level of perceived stress. A moderate stress level is considered between 20-25 points, and a high stress level is considered when obtaining >25 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico